CLINICAL TRIAL: NCT02690233
Title: Perioperative Endothelial Dysfunction in Patients Undergoing Minor Abdominal Surgery. The POETRY Minor Study.
Brief Title: Perioperative Endothelial Dysfunction in Patients Undergoing Minor Abdominal Surgery
Acronym: POETRYminor
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Victoria Ekeløf Busch, MD, Zealand University Hospital
Other Study IDs: POETRY minor
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Injury
Keywords: endothelial dysfunction; surgery; cardiovascular complications; EndoPat; myocardial injury; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood will be collected from a larger vein (e.g. the cubital vein).
  Tetrahydrobiopterin: Blood is sampled into 4mL EDTA tubes. Immediately after withdrawal, a minimum of 1mL blood is mixed with 25μL DTE. The mixture is centrifuged at 2000g for 5 minutes. Plasma is frozen and stored at -80°C.
  Arginine and ADMA: Blood is sampled into 4mL EDTA tubes. Blood samples will be centrifuged at 3000g for 10 minutes, plasma frozen and stored at -80°C until analyzed with high performance liquid chromatography.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Elective Surgery — Elective laparoscopic inguinal hernia repair

SUMMARY:
This study on minor surgery serves to explore whether a dose-response relationship exists between surgical stress and endothelial dysfunction in the early postoperative period. The aim of this explorative and observational clinical study is to closely examine the endothelial function and its dynamics in the early postoperative period after minor surgery (lap. inguinal hernia repair). The endothelial function will be assessed indirectly by EndoPat and plasma biomarkers of nitric oxide bioavailability. The study will contribute to the understanding of perioperative myocardial injury, which is crucial for optimized treatment of patients at risk of cardiovascular complications.

DETAILED DESCRIPTION:
The investigators will include 60 patients undergoing elective inguinal hernia repair. The endothelial function will be measured before surgery and 4 hours after surgery with the EndoPat system. The NO-bioavailibility will be measured by plasma l-arginine, plasma ADMA and plasma biopterins.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a laparoscopic inguinal hernia repair
* Patients ≥ 18 years old

Exclusion Criteria:

* Not capable of giving informed consent after oral and written information
* Previously included in the trial ￼￼ - Surgery within 7 days of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators expect that minor surgery will reduce the reactive hyperemia index assessed 4 hours postoperatively with 15% equal to 1.59. With a power of 0.80 and α on 0.05, the investigators will need to include 54 patients in this study. In order to improve the power of the study, the investigators will include a total of 60 patients.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function assessed by the EndoPat system | At baseline and 4 hours postoperatively

SECONDARY OUTCOMES:
Change in biomarkers of endothelial function: plasma arginine, plasma ADMA, plasma biopterins | At baseline and 4 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sarah VE Busch, MD, Principal Investigator — Department of Surgery, Køge Hospital
Locations (1):
- Department of Surgery, Koge Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devereaux PJ, Goldman L, Cook DJ, Gilbert K, Leslie K, Guyatt GH. Perioperative cardiac events in patients undergoing noncardiac surgery: a review of the magnitude of the problem, the pathophysiology of the events and methods to estimate and communicate risk. CMAJ. 2005 Sep 13;173(6):627-34. doi: 10.1503/cmaj.050011. PMID 16157727
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Landesberg G, Beattie WS, Mosseri M, Jaffe AS, Alpert JS. Perioperative myocardial infarction. Circulation. 2009 Jun 9;119(22):2936-44. doi: 10.1161/CIRCULATIONAHA.108.828228. No abstract available. PMID 19506125
- [Background] Widlansky ME, Gokce N, Keaney JF Jr, Vita JA. The clinical implications of endothelial dysfunction. J Am Coll Cardiol. 2003 Oct 1;42(7):1149-60. doi: 10.1016/s0735-1097(03)00994-x. PMID 14522472
- [Background] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Background] Munzel T, Sinning C, Post F, Warnholtz A, Schulz E. Pathophysiology, diagnosis and prognostic implications of endothelial dysfunction. Ann Med. 2008;40(3):180-96. doi: 10.1080/07853890701854702. PMID 18382884
- [Background] Hu YJ, Wei AN, Chook P, Yin Y, Cheng W, Wu MJ, Celermajer DS, Woo KS. Impact of non-cardiovascular surgery on reactive hyperaemia and arterial endothelial function. Clin Exp Pharmacol Physiol. 2013 Jul;40(7):466-72. doi: 10.1111/1440-1681.12111. PMID 23662794
- [Background] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Menzoian JO, Vita JA. Risk stratification for postoperative cardiovascular events via noninvasive assessment of endothelial function: a prospective study. Circulation. 2002 Apr 2;105(13):1567-72. doi: 10.1161/01.cir.0000012543.55874.47. PMID 11927524
- [Background] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Nedeljkovic ZS, Menzoian JO, Vita JA. Predictive value of noninvasively determined endothelial dysfunction for long-term cardiovascular events in patients with peripheral vascular disease. J Am Coll Cardiol. 2003 May 21;41(10):1769-75. doi: 10.1016/s0735-1097(03)00333-4. PMID 12767663
- [Background] McIlroy DR, Chan MT, Wallace SK, Symons JA, Koo EG, Chu LC, Myles PS. Automated preoperative assessment of endothelial dysfunction and risk stratification for perioperative myocardial injury in patients undergoing non-cardiac surgery. Br J Anaesth. 2014 Jan;112(1):47-56. doi: 10.1093/bja/aet354. Epub 2013 Oct 29. PMID 24172055
- [Background] Hamburg NM, Benjamin EJ. Assessment of endothelial function using digital pulse amplitude tonometry. Trends Cardiovasc Med. 2009 Jan;19(1):6-11. doi: 10.1016/j.tcm.2009.03.001. PMID 19467447
- [Background] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Derived] Ekeloef S, Godthaab C, Schou-Pedersen AMV, Lykkesfeldt J, Gogenur I. Peri-operative endothelial dysfunction in patients undergoing minor abdominal surgery: An observational study. Eur J Anaesthesiol. 2019 Feb;36(2):130-134. doi: 10.1097/EJA.0000000000000935. PMID 30543557